CLINICAL TRIAL: NCT06736756
Title: Impact of Tensor Fascia Lata Stretch Prior to Squat on Vastus Medialis Obliqus Activity in Patellofemoral Pain Syndrome
Brief Title: Impact of Tensor Fascia Lata Stretch on Vastus Medialis Obliqus Activity
Status: Recruiting | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Tasneem Khaled Fouad Abdelghany, Teaching Assistant Orthopedic department, Ahram Canadian University
Other Study IDs: Patellofemoral Pain syndrome
Record Dates: First submitted 2024-12-07; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Plyometric Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stretch Exercise — To stretch Tensor fascia lata muscle,each participant starts with side lying position with the tested limb upmost. The lower limb (non-tested) is kept in hip and knee flexion to ensure stability. The tested limb is then taken into hip extension and adduction with knee extended. The exercise is held for 60 seconds and repeated 5 times with 10 seconds break intervals.

SUMMARY:
Patellofemoral pain syndrome (PFPS) is one of the most typical causes of anterior knee pain in adolescents and young adults under the age of 50.It is believed that imbalanced action between quadriceps components, is the most contributing cause of PFPS.Investigating exercises that increase VMO muscle activation and enhance the ratio between VMO and VL have been a standardized target in literature.

DETAILED DESCRIPTION:
Participants will have the assessed limb ready by shaving the hair on thigh and using alcohol swabs to clean the area from any residues.

For the VMO, a surface EMG electrode will be placed 4 cm superior and 4 cm medial to the supromedial boarder of patella at approximately 55 degrees to the long axis of the femur. As for the VL, the electrode will be placed 10 cm superior and 6-8 cm lateral to the superior lateral boarder of the patella and orientated 15 degrees to the vertical. All electrodes are self-adhesive (Figure 8) and will be connected to EMG sensors that will be attached and secured by double-sided tape.Each participant will perform three consecutive squats with 5 seconds interval break between each repetition. The squat depth will be kept at 50 degrees knee flexion. Mean muscle activity from three squat repetitions of VMO and VL is recorded and VMO:VL ratio is calculated. Afterward, each participant will perform the TFL stretch and repeat the three squats again.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders.
2. Body mass index (BMI) ranges from 18.5 to 29.9.
3. Age ranges between 18 and 30 years old.
4. Experience nontraumatic anterior knee pain.
5. Pain with any two activities, including running, jumping, squatting, kneeling, stair ascent/descent or prolonged sitting.
6. Having at least one positive PFPS clinical tests including, patellofemoral compression, patellofemoral gliding or resistive quadriceps setting

Exclusion Criteria:

1. Coexisting pathology around the knee, including patellar subluxation or dislocation.
2. Previous knee surgery.
3. Suspicion of patellar tendinopathy, with strong consideration of pain localised to the patellar tendon.
4. Patients didn't receive physiotherapy treatment or use of non-steroidal anti-inflammatory drugs for knee pain in the previous 3 months.
5. Any neurological or rheumatic disorders
6. Pain intensity more than 5 (based on visual analogue scale)
7. Hip and ankle pathology.
8. BMI more than 30%.
9. Pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients referred from orthopedic surgeon with diagnosis of PFPS
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
VMO muscle activity | During the procedure
  VMO muscle activity during squat is assessed by EMG device

SECONDARY OUTCOMES:
VMO to VL ratio | Immediately after the procedure
  Ratio between VMO and VL activity during squat

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy, Professor, Principal Investigator — Cairo University
Locations (1):
- Tasneem Khaled, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No